CLINICAL TRIAL: NCT05660629
Title: Comparison of the Effects of Exercise and Protective Approach in the Rheumatoid Hand and Joint Mobilization Applications on Pain, Functional Status and Quality of Life
Brief Title: Mulligan Mobilization in Rheumatoid Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ahi Evran University
Record Dates: First submitted 2022-11-30; First posted 2022-12-21 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Mulligan Mobilization; Hand Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mulligan Mobilization (Experimental): Rehabilitation Program (Active wrist ROM exercises):
  * Forearm pronation and supination
  * Wrist flexion and extension
  * Wrist flexion and extension (in the form of a fist)
  * MCP Joint Flexion and Extension
  * Thumb IC joint Flexion and Extension
  * Abduction and Adduction of Fingers
  These exercises will be performed by the physiotherapist in the form of 5 seconds of movement / 15 seconds of rest, 10 repetitions a day, 5 days a week for 6 weeks.
  Mulligan Mobilization:
  * Carpal Medio-lateral Glide (open kinetics, wrist flexion and extension movement)
  * Carpal Rotation (open kinetics, wrist flexion and extension)
  * Scaphoid Antero-posterior Glide (open kinetics)
  * Metacarpal Antero-posterior Glide (When Clenching)
  * Medio-lateral Glide to PIP-DIP joints (open kinetics, fingers flexed)
  Interventions: Other: Mulligan Mobilization
- Sham Mobilization (Sham Comparator): Participants will receive sham mobilization in addition to the ROM exercises given in the Mulligan group. Sham mobilization will be done in the same position as Mulligan but without any glide force.
  Interventions: Other: Mulligan Mobilization
- Control (No Intervention): Participants will receive therapeutic patient training consisting of home exercise recommendations, basic disease information, physical activity advice, and joint protection methods.

INTERVENTIONS:
Other: Mulligan Mobilization — Mobilization with movement (MWM) is the concurrent application of sustained accessory mobilization applied by a therapist and an active physiological movement to end range applied by the patient. Passive end-of-range overpressure, or stretching, is then delivered without pain as a barrier.
  Arms: Mulligan Mobilization; Sham Mobilization

SUMMARY:
The goal of this randomized-controlled study is to learn about the effectiveness of the Mulligan mobilization in rheumatoid hands. The main question it aims to answer are:

-Does mulligan mobilization reduce effusion in wrist joints with rheumatoid arthritis? Participants will take Mulligan mobilization application and active ROM exercises for their hands. Researcher will compare treatments group ith sham mobilization.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic disease that can lead to chronic pain, bone and soft tissue damage, and disability retirement. Alleviating pain and maintaining joint range of motion in RA are important for reducing disability. Joint mobilizations are manual therapy techniques used to increase range of motion and reduce pain. The aim of this study is to investigate the effects of rheumatoid hand exercise and protective approach and joint mobilization applications on pain, functional status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with RAS according to ACR and EULAR criteria,
* Being under the control of a physiatrist for at least 1 year,
* Have not had any upper extremity surgery in the last 6 months
* Have the cognitive capacity to understand commands,
* Not to be involved in any other rehabilitation program or study,

Exclusion Criteria:

* Presence of soft tissue injury and chronic bone damage in the hand,
* Presence of acute inflammation in any joint in the previous week,
* Presence of a degenerative or non-degenerative neurological condition that causes a change in pain perception,

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Joint activity | 6 weeks
  Primary outcomes included the automated quantification (Q) of joint activity using color Doppler pixel count calculations (% hyperemia/blood flow activity score within an inflamed joint: color Q-Doppler MCP/region)
Amount of hypertrophia and effusion in wrist joints | 6 weeks
  Synovial fluid (area of hypertrophy and effusion, mm2: synovial fluid MCP/region)
Distance in wrist joints | 6 weeks
  the radiographic distance (mm) between the MCP or interphalangeal bone space (joint space MCP/region)
DAS-28 | 6 weeks
  High disease activ ity >5.1, low disease activity ≤ 3.2, remission ≤ 2.6

SECONDARY OUTCOMES:
Determining the state of pain after treatment | 6 weeks
  Pain will be assessed using the Mcgill-Melzack Pain Questionnaire
Grip force | 6 weeks
  Hand grip strength will be measured with a pinch meter and a dynamometer
Range of Motion | 6 weeks
  Range of Motion will be measured with goniometer
Post-treatment status of disease-related quality of life | 6 weeks
  Quality of life was assessed using the Rheumatoid Arthritis Quality of Life (RAQoL).
Physical, social, and emotional well-being in RA | 6 weeks
  Arthritis Impact Measurement Scales (AIMS)

CONTACTS AND LOCATIONS:
Overall Officials: Figen TUNCAY, Professor, Study Director — Kirsehir Ahi Evran Universitesi
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data will be done using the Google Drive link.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: It will be shared for 2 years.

REFERENCES:
- [Result] Levitsky A, Kisten Y, Lind S, Nordstrom P, Hultholm H, Lyander J, Hammelin V, Gentline C, Giannakou I, Faustini F, Skillgate E, van Vollenhoven R, Sundberg T. Joint Mobilization of the Hands of Patients With Rheumatoid Arthritis: Results From an Assessor-Blinded, Randomized Crossover Trial. J Manipulative Physiol Ther. 2019 Jan;42(1):34-46. doi: 10.1016/j.jmpt.2018.04.007. Epub 2019 Mar 14. PMID 30879707
- [Result] Villafane JH, Cleland JA, Fernandez-de-Las-Penas C. Bilateral sensory effects of unilateral passive accessory mobilization in patients with thumb carpometacarpal osteoarthritis. J Manipulative Physiol Ther. 2013 May;36(4):232-7. doi: 10.1016/j.jmpt.2013.05.008. Epub 2013 May 27. PMID 23719518
- [Result] Ozcelep OF, Ustun I, Algun ZC. Effect of task-oriented training on pain, functionality, and quality of life in rheumatoid arthritis. Turk J Phys Med Rehabil. 2022 Mar 1;68(1):76-83. doi: 10.5606/tftrd.2022.6666. eCollection 2022 Mar. PMID 35949976
- [Derived] Ozcelep OF, Tunali N, Turhan A, Polat E, Demir C, Gumusay D, Tuncay F. The effect of mobilization with movement on pain, joint distance, effusion area, and inflammation in rheumatoid arthritis: a double-blind randomized controlled clinical trial. J Orthop Surg Res. 2025 Oct 28;20(1):929. doi: 10.1186/s13018-025-06121-3. PMID 41152887